CLINICAL TRIAL: NCT02709330
Title: An Open-label, Single-center, 12-month Trial of a Lunasin Regimen for Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: ALS Reversals - Lunasin Regimen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Richard Bedlack, M.D., Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Richard Bedlack, M.D., Ph.D., Associate Professor of Neurology, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00063754
Record Dates: First submitted 2016-03-05; First posted 2016-03-16 (Estimated); Results first posted 2018-12-13 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-11

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Historically Controlled Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lunasin regimen (Experimental): The Lunasin regimen consists of:
  * LunaRich X Capsules (12 capsules per day)
  * Reliv NOW - a mixture of 'vitamins, minerals and super-powered antioxidants' (3 scoops per day)
  * Pro-Vantage - a mixture of 'soy protein, medium chain triglycerides, creatine, CoQ10 and supercharged amino acids' (2 scoops per day)
  It will be suggested that patients open the LunaRich X capsules and mix the contents of these as well as the other 2 ingredients in water to make a shake. If patients do not tolerate advancing to the next dosage, they will be asked to drop back to the highest dosage they could tolerate.
  Interventions: Drug: Lunasin Regimen
- Historical controls (Active Comparator): For each enrolled participant, matched historical controls will be identified from the PatientsLikeMe database. Participants will be matched according to their ALSFRS-R progression rate before they start on the Lunasin regimen (estimated by assuming their score was normal at 48 on the date of symptom onset).
  Interventions: Other: Historical control

INTERVENTIONS:
Drug: Lunasin Regimen — LunaRich X Capsules, Reliv Now, ProVantage
  Arms: Lunasin regimen
Other: Historical control — Matched historical controls will be identified from the PatientsLikeMe database.
  Arms: Historical controls

SUMMARY:
This is a 12-month, widely inclusive, largely virtual, single-center, open-label pilot trial utilizing a historical control group. Participants will receive a Lunasin regimen and will be asked to register for an account of PatientsLikeMe website, where after the initial in-clinic visit, they will be asked to enter specific data.

DETAILED DESCRIPTION:
The primary hypothesis is that a supplement regimen containing Lunasin (referred to as the Lunasin regimen) can decrease the rate of ALSFRS-S progression by 50% relative to matched historic controls.

ALS is a devastating motor neuron disease that causes rapidly progressive muscle weakness, disability and premature death. In spite of a large number of attempted ALS trials, there are no significant disease-modifying therapies for this condition.

It was recently reported that a patient with a validated diagnosis of ALS, had experienced dramatic objective improvement in speech, swallowing and limb strength while taking a supplement regimen containing Lunasin. Several other patients with ALS have also reported improvement on this Lunasin regiment, though records were not obtainable to validate these.

The Lunasin regimen will consist of:

* LunaRich X Capsules
* Reliv NOW - a mixture of 'vitamins, minerals and super-powered antioxidants'
* Pro-Vantage - a mixture of 'soy protein, medium chain triglycerides, creatine, CoQ10 and supercharged amino acids'

Dosages will be titrated up to target over the first 6 days. The subject will take the highest tolerated dosing for the remainder of the 12-month study.

There are 3 in-clinic visits which occur at screening/baseline, Month 1 and Month 12. For Months 2-11, participants will make "virtual visits" by measuring their own ALSFRS-R score and weight and will record it in the PatientsLikeMe website. They will also self-report any perceived efficacy, compliance, adverse events and changes in concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged at least 18 years.
* Sporadic or familial ALS diagnosed as possible, laboratory-supported probable, probable, or definite as defined by revised El Escorial criteria.
* Patient is able to understand and express informed consent (in the opinion of the site investigator).
* Patient has access to the Internet on a desktop computer, laptop, or tablet and has a working email address.
* Patient or caregiver is willing and able to use a computer and enter data on a secure website.
* Patient is able to read and write English.
* Women must not be able to become pregnant (e.g., post-menopausal, surgically sterile, or using adequate birth control methods) for the duration of the study and three months after study completion. Adequate contraception includes: abstinence, hormonal contraception (oral contraception, implanted contraception, injected contraception or other hormonal contraception, for example patch or contraceptive ring), intrauterine device (IUD) in place for ≥ 3 months, barrier method in conjunction with spermicide, or another adequate method.

Exclusion Criteria:

* Patient is taking other experimental treatments for ALS.
* Prior side effects from Lunasin.
* Known soy allergy.
* Patient has a medical or psychiatric illness that could in the investigator's opinion interfere with the patient's ability to participate in this study.
* Pregnant women or women currently breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-09-13 (Actual); Study Completion 2017-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bedlack, M.D., Ph.D., Principal Investigator — Associate Professor of Neurology
Locations (1):
- Duke Medicine / Neurology, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants will be assigned a global unique ID number (GUID), which will allow de-identified data sharing.

REFERENCES:
- [Derived] Bedlack RS, Wicks P, Vaughan T, Opie A, Blum R, Dios A, Sadri-Vakili G. Lunasin does not slow ALS progression: results of an open-label, single-center, hybrid-virtual 12-month trial. Amyotroph Lateral Scler Frontotemporal Degener. 2019 May;20(3-4):285-293. doi: 10.1080/21678421.2018.1556698. Epub 2019 Jan 21. PMID 30663902

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the clinic patient population and outside advertisements and postings. Recruitment began 3/28/2016 and ended 9/14/16 once 50 subjects had been enrolled. Study visits were conducted at the Duke ALS clinic and via phone contacts.
Pre-assignment Details: An additional 10 subjects were consented specifically as controls for outcome measure 2 and not included in the treatment group (Lunasin regimen).
Groups:
- Lunasin Regimen: The Lunasin regimen consists of:
  * LunaRich X Capsules (12 capsules per day)
  * Reliv NOW - a mixture of 'vitamins, minerals and super-powered antioxidants' (3 scoops per day)
  * Pro-Vantage - a mixture of 'soy protein, medium chain triglycerides, creatine, CoQ10 and supercharged amino acids' (2 scoops per day)
  It will be suggested that patients open the LunaRich X capsules and mix the contents of these as well as the other 2 ingredients in water to make a shake. If patients do not tolerate advancing to the next dosage, they will be asked to drop back to the highest dosage they could tolerate.
  Lunasin Regimen: LunaRich X Capsules, Reliv Now, ProVantage
- Control: Subjects were consented specifically as controls for outcome measure 2 and not included in the treatment (Lunasin regimen) group.
Period: Overall Study
Arm/Group | Lunasin Regimen | Control
Started | 50 | 10
Completed | 37 | 10
Not Completed | 13 | 0
Not completed — Death | 5 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 4 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data were not collected for the 5 ALS control subjects and 5 healthy control subjects.
Arm/Group | Lunasin Regimen
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 47
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Change in Revised ALS Functional Rating Scale (ALSFRS-R)
Description: ALSFRS-R is a quickly administered (five minute) ordinal rating scale used to determine patient's assessment of their capability and independence in 13 functional activities. All 13 activities are relevant in ALS. Each task is rated on a five-point scale from 0 = can't do, to 4 = normal ability, with a total score of 52 points. Reported is the rate of change in total points per month.
Time Frame: Screening/baseline - 12 months
Population: 1 participant deleted PLM account; 2 others did not enter ALSFRS-R data.
Measure: Mean (Standard Deviation); unit: points per month
Arm/Group | Lunasin Regimen
Number analyzed (Participants) | 47
points per month | 0.44 (1.6)
Statistical Analysis 1: Comparison: Lunasin Regimen; Matched historical controls will be identified from the PatientsLikeMe database; Test type: Other; p = 0.99, Kolmogorov-Smirnov Test

2. Secondary Outcome: Change in H3 Histone Acetylation
Description: Participants, ALS controls (not on Lunasin) and healthy controls (not on Lunasin) had blood drawn at baseline and 1 month time points. Histones were extracted from blood cells. Western blots were used to look at specific histone acetylation patterns that Lunasin had reportedly altered in cell cultures (H3K9K14ac2 and H4K5K8K12K16). Integrated density values for AcH3 protein bands were normalized for total H3. Percent H3 values for the 1 month time point were normalized to that of the baseline visit. Results were analyzed by one-way ANOVA.
Time Frame: Screening/baseline, Month 1
Population: Lunasin regimen: 20 of 50 enrolled participants did not have sufficient sample. Five ALS control subjects (not on Lunasin) and five healthy control subjects (not on Lunasin) were also consented specifically for this analysis. One of the healthy controls did not have sufficient sample.
Measure: Mean (Standard Deviation); unit: percentage of baseline
Groups:
- ALS Controls: Individuals with ALS who are not on Lunasin.
- Healthy Controls: Healthy individuals who are not on Lunasin.
Arm/Group | Lunasin Regimen | ALS Controls | Healthy Controls
Number analyzed (Participants) | 30 | 5 | 4
percentage of baseline | 0.993 (0.53) | 1.252 (0.74) | 1.795 (1.29)
Statistical Analysis 1: Comparison: Lunasin Regimen vs ALS Controls vs Healthy Controls; Test type: Other; p = 0.0748, ANOVA

3. Secondary Outcome: Percent Agreement Between the Weights Obtained by Patients and Study Coordinator
Description: To confirm that participants can accurately measure their own weight, even as they become more disabled by ALS, the investigators will compare the participant-generated weight with the weight obtained by the study coordinator at the Month 1 and Month 12 visits. A simple description of the accuracy (percent agreement between the weights) will be used.
Time Frame: Month 1, Month 12
Population: Participants with both self-obtained weight and weight obtained by the study coordinator available.
Measure: Number (95% Confidence Interval); unit: percentage of agreement
Arm/Group | Lunasin Regimen
Number analyzed (Participants) | 49
percentage of agreement
  Month 1 | 99.47 [99.07 to 99.70]
  Month 12: number analyzed (Participants) | 25
  Month 12 | 99.05 [94.28 to 99.58]
Statistical Analysis 1: Comparison: Lunasin Regimen; Test type: Other; p < 0.00001, Lin's Concordance

4. Secondary Outcome: Enrollment Rate
Description: Rate of enrollment in reaching the 50 participants required to fill the trial.
Time Frame: Screening/baseline - Month 12
Measure: Number; unit: participants per month
Arm/Group | Lunasin Regimen
Number analyzed (Participants) | 50
participants per month | 9.1

5. Secondary Outcome: Retention Rate
Description: Percentage of surviving participants who completed the month 12 visit.
Time Frame: Month 12
Measure: Number; unit: percentage of participants
Arm/Group | Lunasin Regimen
Number analyzed (Participants) | 50
percentage of participants | 84

6. Secondary Outcome: Frequency of ALS Reversals
Description: The percentage of enrolled participants experiencing an ALSFRS-R improvement of at least 4 points lasting at least 12 months.
Time Frame: Screening/baseline - Month 12
Measure: Number; unit: percentage of participants
Arm/Group | Lunasin Regimen
Number analyzed (Participants) | 50
percentage of participants | 0

7. Secondary Outcome: ALSFRS-R Accuracy
Description: To confirm that participants can accurately measure their own ALS Functional Rating Scale (Revised, ALSFRS-R), the investigators will compare the ALSFRS-R obtained by the coordinator with that obtained by the participants themselves at the Month 1 Visit. Correlational analysis between these 2 scores will be performed with Spearman's rho.
Time Frame: Month 1
Population: 2 participants did not provide month 1 scores.
Measure: Mean (95% Confidence Interval); unit: percentage of accuracy
Arm/Group | Lunasin Regimen
Number analyzed (Participants) | 48
percentage of accuracy | 99.39 [98.92 to 99.65]
Statistical Analysis 1: Comparison: Lunasin Regimen; Test type: Other; p < 0.00001, Lin's Concordance

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse Event data were not collected for the 5 ALS control subjects and 5 healthy control subjects.
Arm/Group | Lunasin Regimen
All-Cause Mortality (participants affected / at risk) | 5/50
Serious Adverse Events (participants affected / at risk) | 13/50
Other Adverse Events (participants affected / at risk) | 45/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lunasin Regimen (N=50)
Death from ALS progression (Nervous system disorders) | 3
Death from Intracerebral Hemorrhage (Nervous system disorders) | 1
Death from Cardiac Arrest (Cardiac disorders) | 1
Obstipation/Fecal Imaction (Gastrointestinal disorders) | 2
Intracerebral Hemorrhage (Nervous system disorders) | 1
PEG Infection (Infections and infestations) | 1
Subdural Hematoma (Nervous system disorders) | 1
C. Diff Infection (Infections and infestations) | 1
Mumps Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Cardiac Arrest (Cardiac disorders) | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lunasin Regimen (N=50)
Constipation (Gastrointestinal disorders) | 11
Fullness/early satiety (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 3
Decreased Appetite (Gastrointestinal disorders) | 2
Increased ALS progression (Nervous system disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Itching (Skin and subcutaneous tissue disorders) | 2
Carbon Dioxide Retention (Respiratory, thoracic and mediastinal disorders) | 1
Hand and Finger Swelling (Musculoskeletal and connective tissue disorders) | 1
Increased Appetite (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Hyperglycemia (Endocrine disorders) | 1
Irritated Hiatal Hernia (Musculoskeletal and connective tissue disorders) | 1
Fall (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
Worsened Anxiety (Psychiatric disorders) | 1
Prostate Enlargement (Renal and urinary disorders) | 1
Restless Arm Movements (Nervous system disorders) | 1
Increased Fasciculations (Nervous system disorders) | 1
UTI (Infections and infestations) | 1
Increased Cramps (Nervous system disorders) | 1
Increased Pseudobulbar Affect (Nervous system disorders) | 1
Breast Tenderness (Musculoskeletal and connective tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Heaviness (Nervous system disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Hyponatremia (Blood and lymphatic system disorders) | 1
Ear Ache (Musculoskeletal and connective tissue disorders) | 1
Weight Gain (Gastrointestinal disorders) | 1
Weight Loss (Gastrointestinal disorders) | 1
Influenza Infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT02709330/Prot_SAP_000.pdf